CLINICAL TRIAL: NCT01306383
Title: Assessment of the Health Benefits Associated With Consumption of Solar Disinfection of Drinking Water by Children Under Age 5 Years, With Particular Emphasis on Dysentery and Childhood Diarrhoea
Brief Title: Solar Disinfection (SODIS) of Drinking Water for Use in Developing Countries or in Emergency Situations
Acronym: SODISWATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: ICROSS, Kenya (Unknown); International Water and Sanitation Development (IWSD), Zimbabwe (Unknown); CARE International - Cambodia (CIC), Cambodia (Unknown)
Responsible Party: Dr Kevin McGuigan PhD BSc FInstP / Project Coordinator, Royal College of Surgeons in Ireland (RCSI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SODISWATER EU 031650; SODIS Kenya, Zimbab, Cambodia (Other: EU 031650)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-02

CONDITIONS: Dysentery; Diarrhoea
Keywords: SODIS; waterborne; Disease; Diarrhoea; dysentery
MeSH Terms: conditions — Dysentery; Diarrhea; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SODIS Bottles given (Active Comparator): Caregivers in the intervention group were given two 2-litre plastic bottles. Bottle was filled with available water and placed in direct sunlight for a minimum of 6 hours. Water was consumed the next day while second bottle was being consumed.
  Interventions: Other: SODIS Bottle
- Usual practices (Active Comparator): Caregivers in this group were asked to maintain their usual practices regarding drinking water so that disease rates could be compared with the SODIS arm
  Interventions: Other: SODIS Bottle

INTERVENTIONS:
Other: SODIS Bottle — SODIS Bottles used by SODIS group to treat their drinking water
  Other Names: Unused 2-litre PET bottles (e.g. Coca-Cola, Pepsi)

SUMMARY:
SODISWATER was a health impact assessment study investigating the effect of sunlight to inactivate microbial pathogens in drinking water. This study was carried out by observing whether children younger than 5 years old who drink solar disinfected water were healthier than those who did not. Health was measured by how often the children had diarrhoea or dysentery.

Caregivers for the participants were given plastic bottles to place in the sun, water samples were then collected from these plastic bottles to be analyzed. They were also requested to fill in diarrhea diaries.

TESTABLE RESEARCH HYPOTHESES:

Health Impact Assessment: Children who use solar disinfected water will have:

(a) lower morbidity due to non-bloody diarrhoea and bloody diarrhoea (c) increased growth rates (d) lower mortality (e) increased family productivity (f) decreased care-giver burden (g) increased school attendance

DETAILED DESCRIPTION:
The current evidence base for solar disinfection in the prevention of diarrhoeal disease in children rests on three published studies. All share two significant weaknesses: all were carried out in Kenya, in communities which have very high incidences of diarrhoeal disease and water characterised by high levels of both turbidity and microbial contamination. Furthermore, neither of the studies of diarrhoeal disease distinguished between dysentery (associated with significant risk of mortality) and other sorts of diarrhoea, which carry a far lower risk. The present study will extend the evidence base into communities at lower risk and with higher water quality. Furthermore, by using pictorial diaries, dysentery can be analysed as a specific health endpoint. Diarrhoea will be recorded consistent with the World Health organisation definition: three or more loose or watery stools in a 24-hour period and/or stools containing blood or mucus.

AIM OF THE PROJECT IN RELATION TO HEALTH IMPACT ASSESSMENT STUDIES:

The primary aim of the SODISWATER PROJECT is to demonstrate that SODIS is an appropriate intervention against diarrhoeal and waterborne disease among communities in developing countries and those affected by natural or man-made disasters by conducting multi-centred epidemiologically controlled Health Impact Assessments of the SODIS technique across the African Continent under a variety of social, geographical and climactic conditions.

SCIENTIFIC OBJECTIVES OF SODISWATER IN RELATION TO HEALTH IMPACT ASSESSMENT STUDIES:

1. Assessment of the change in health reasonably attributed to the provision of solar disinfected drinking water at the point of use in 3 countries (Kenya, Zimbabwe and Cambodia).
2. Assessment of the relationship between solar disinfected drinking water and selected health indicators (including morbidity due to non-bloody diarrhoea and dysentery, weight loss, mortality, growth rates, productivity, care-giver burden, and school attendance. Mortality will also be monitored but the sample sizes are of insufficient size to produce detailed information and scaling up, to account for this is not possible due to prohibitive costs).
3. Demonstration of the effectiveness of SODIS at household level.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more children aged less than 5 years in the household

Exclusion Criteria:

* Chlorinated piped water source available in household

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Dysentery disease rate | 12 month
  Incidence of occurrence of blood or mucous in diarrhoeal stools was noted by caregivers and recorded in a pictorial diary which was collected every 2 weeks.
Diarrhoea disease rate | 12 months
  Incidence of diarrhoea and numbers of diarrhoeal episodes was noted by caregivers and recorded in a pictorial diary which was collected every 2 weeks.

SECONDARY OUTCOMES:
Height and weight benefit | 12 months
  Anthropometric measurements of height and weight were recorded at 3 month intervals across the 12 month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G McGuigan, PhD, Principal Investigator — RCSI
Locations (3):
- CIC, Phnom Penh, Phnom Penh, Cambodia
- ICROSS, Nairobi, Ngong Hills, Kenya
- IWSD, Harare, Mount Pleasant, Zimbabwe

REFERENCES:
- [Background] Du Preez M, Mcguigan KG, Conroy RM. Solar disinfection of drinking water in the prevention of dysentery in South African children aged under 5 years: the role of participant motivation. Environ Sci Technol. 2010 Nov 15;44(22):8744-9. doi: 10.1021/es103328j. PMID 20977257
- [Background] Ubomba-Jaswa E, Fernandez-Ibanez P, McGuigan KG. A preliminary Ames fluctuation assay assessment of the genotoxicity of drinking water that has been solar disinfected in polyethylene terephthalate (PET) bottles. J Water Health. 2010 Dec;8(4):712-9. doi: 10.2166/wh.2010.136. Epub 2010 Apr 13. PMID 20705982
- [Background] Conroy RM, Meegan ME, Joyce T, McGuigan K, Barnes J. Solar disinfection of drinking water protects against cholera in children under 6 years of age. Arch Dis Child. 2001 Oct;85(4):293-5. doi: 10.1136/adc.85.4.293. PMID 11567937
- [Background] Conroy RM, Elmore-Meegan M, Joyce T, McGuigan KG, Barnes J. Solar disinfection of drinking water and diarrhoea in Maasai children: a controlled field trial. Lancet. 1996 Dec 21-28;348(9043):1695-7. doi: 10.1016/S0140-6736(96)02309-4. PMID 8973432
- [Derived] du Preez M, Conroy RM, Ligondo S, Hennessy J, Elmore-Meegan M, Soita A, McGuigan KG. Randomized intervention study of solar disinfection of drinking water in the prevention of dysentery in Kenyan children aged under 5 years. Environ Sci Technol. 2011 Nov 1;45(21):9315-23. doi: 10.1021/es2018835. Epub 2011 Oct 5. PMID 21936492
- See also: SODISWATER project website — http://www.rcsi.ie/sodis
- See also: Information site for SODIS — http://www.sodis.ch